CLINICAL TRIAL: NCT04793009
Title: Prophylactic Funnel Mesh to Prevent Parastomal Hernia in Permanent End Colostomy: A Retrospective Cohort Study
Brief Title: Prophylactic Funnel Mesh to Prevent Parastomal Hernia in Permanent End Colostomy After Abdomino-perineal Resection
Status: Completed | Type: Observational
Sponsor: Walter Brunner (Other)
Responsible Party: Sponsor-Investigator, Walter Brunner, Leitender Arzt kolorektale Chirurgie, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Other Study IDs: CHIR2021WB; 2021-00120 (Other: BASEC)
Record Dates: First submitted 2021-03-01; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Hernia; Colostomy Stoma
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- mesh group: patients undergoing abdominoperineal resection with end colostomy and implantation of a prophylactic, funnel-shaped, intraperitoneal mesh
  Interventions: Device: funnel-shaped, intraperitoneal mesh placement
- no-mesh group: patients undergoing abdominoperineal resection with end colostomy without implantation of a prophylactic, funnel-shaped, intraperitoneal mesh

INTERVENTIONS:
Device: funnel-shaped, intraperitoneal mesh placement — Implantation of a prophylactic, 3D funnel-shaped, intraperitoneal, non-absorbable and synthetic mesh (Dyna Mesh IPST 2x15x15 cm™ and 3x16x16 cm™, FEG Textiltechnik, Aachen, Germany,)
  Groups: mesh group

SUMMARY:
This retrospective study asses if a prophylactic, funnel-shaped, intraperitoneal mesh prevents parastomal hernia in patients undergoing abdominoperineal rectum resection with permanent end colostomy.

ELIGIBILITY:
Inclusion Criteria:

* elecitve abdominoperineal resection

Exclusion Criteria:

* rejection of a retrospective data Analysis
* age under 18 years
* meshes other than the funnel-shaped mesh

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving elective abdominoperineal resection between January 2013 and December 2018 at the Cantonal Hospital of St. Gallen
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Occurrence of parastomal hernia | initial operation until an avarage of 3 years
  clinical or radiological diagnosed parastomal hernia

SECONDARY OUTCOMES:
Reoperations due to parastomal hernia | initial operation until an avarage of 3 years
  Reoperation due to problems caused by parastomal hernia
Mesh-associated complications | initial operation until an avarage of 3 years
  any complications due to the mesh

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available to researchers whose proposed use of the data has been approved.

REFERENCES:
- [Derived] Ammann Y, Widmann B, Sparn M, Warschkow R, Weitzendorfer M, Brunner W. Prophylactic funnel mesh to prevent parastomal hernia in permanent end colostomy: A retrospective cohort study. Colorectal Dis. 2021 Oct;23(10):2627-2636. doi: 10.1111/codi.15817. Epub 2021 Sep 4. PMID 34265151